CLINICAL TRIAL: NCT01515358
Title: A Single-Dose, Dose-Escalation Study to Evaluate the Safety and Tolerability of LY3000328 in Healthy Subjects
Brief Title: A Study to Evaluate the Safety and Tolerability of LY3000328 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 14340; I5U-MC-ANBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY3000328

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Single dose of placebo administered orally in 1 out of 3 study periods separated by at least a 7-day wash-out period between each dose.
  Interventions: Drug: Placebo
- LY3000328 (Experimental): Single escalating dose of up to 300 mg/kg of LY3000328 administered orally in 2 out of 3 study periods separated by at least a 7 day wash-out period between each dose.
  Interventions: Drug: LY3000328

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: LY3000328 — Administered orally
  Arms: LY3000328

SUMMARY:
The purposes of this study are to determine the safety and side effects of LY3000328, to determine how well the body will tolerate LY3000328, and to determine how long LY3000328 remains in the body.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined by medical history and physical examination

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more drug related adverse events (AEs) or any serious AEs | Baseline to study completion (estimate 3 months)

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve (AUC) of LY3000328 | Pre-dose up to Day 6 post-dose
Pharmacokinetics: Maximum concentration (Cmax) of LY3000328 | Pre-dose up to Day 6 post-dose
Change in Cathepsin S (CatS) activity | Pre-dose, up to 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore